CLINICAL TRIAL: NCT04879784
Title: Primary Prevention of Cytomegalovirus in Pregnancy: Addressing the Gaps (CMV GAP)
Acronym: CMV GAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: St George's, University of London (Other); University College, London (Other); St George's University Hospitals NHS Foundation Trust (Other); CMV Action (Unknown); Kingston University (Other); University of Cambridge (Other); University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CHI1088
Record Dates: First submitted 2021-05-07; First posted 2021-05-10 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Cytomegalovirus Congenital
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stored antenatal sera: Antenatal sera from women booking for antenatal care at six centres in England
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
CMV is the most common congenital infection (an infection acquired before birth) in the UK. It is the leading non-genetic cause of sensorineural (inner ear) hearing loss and a common cause of neuro-disability. Congenital CMV is associated with an estimated cost of £732 million each year in the UK.

The risk of acquiring CMV in pregnancy may be reduced by making simple adaptions to behaviours to avoid direct contact with saliva and urine of young children. There are currently no national policies that recommend CMV risk reduction measures in pregnancy.

The overarching aim of project is to establish and build effective partnerships with policy makers and stakeholders to identify policy priorities and to gather the essential evidence required to fully inform policies to reduce the risk of CMV infection in pregnancy.

The specific objective of this element of the overall project is to determine the proportion of women at risk of primary CMV infection in pregnancy and the rates of primary CMV infection in the first trimester of pregnancy by testing blood samples routinely collected at antenatal booking at representative sites in England.

In partnership with University Hospital Southampton NHS Foundation Trust Specialist Virology Laboratory, investigators will carry out a CMV serosurvey using stored antenatal serum from pregnant women across England. Investigators will test these samples at the point at which they would otherwise be destroyed. This will enable investigators to determine the proportion of women who are seronegative, as this is the group that will be enrolled in future intervention studies (both educational and also vaccine studies). This information is required to accurately inform the power calculation for large efficacy studies. This will also allow investigators to determine the proportion of women who acquire CMV in the first trimester of pregnancy - thus demonstrating the consequences of policy inaction.

DETAILED DESCRIPTION:
Ten children are born every day in the UK with congenital cytomegalovirus (CMV) infection. Over half of infants who have symptoms or signs of CMV at birth have moderate to severe long-term impairments such as hearing loss or neurodisability; of those infants who appear well at birth, nearly 1 in 5 have long-term adverse sequalae. The impact on these families is immense, even for those families whose child has normal hearing and development, as the outcomes are often unpredictable at birth. The cost of CMV in the UK is around £732 million each year.

CMV infection in healthy individuals is often asymptomatic or associated with mild flu-like symptoms and therefore the infection may not be diagnosed in pregnancy. If a woman has a primary CMV infection (i.e. never had CMV infection before, termed 'seronegative'), the risk of transmission to the infant is around 32%; the risk is lower in those women who had had CMV infection previously (CMV IgG antibodies present, termed 'seropositive'), in the order of 1%. Acquisition of CMV infection in the first trimester of pregnancy is associated with the highest risk of adverse outcomes for the infant.

The risk of acquiring CMV in pregnancy can be reduced by making simple adaptions to behaviours to avoid direct contact with saliva and urine of young children - who are the most common transmitters of CMV infection to pregnant women. For example: tasting food first and not eating a young child's left-over food; or kissing on the forehead instead of on the lips; handwashing after nappy changes.

Despite CMV being the most common congenital infection and the leading infectious cause of sensorineural hearing loss and neurodisability, it is much less well known than other conditions that occur at a lower frequency, such as Down's Syndrome.

However, the majority of antenatal care providers do not include information about CMV to women alongside information about how to prevent other, much less common conditions, such as toxoplasmosis. There are currently no national policies that recommend CMV risk reduction measures in pregnancy.

Investigators are working with policy makers and other key stakeholders to identify gaps which need to be addressed in future trials of interventions in pregnancy to reduce the risk of CMV in pregnancy and therefore the number of infants born with congenital CMV infection.

In order to inform these discussions and future research studies, investigators need accurate information about the proportion of women in the UK who are seronegative - that have not had CMV before. This is because future studies will enrol seronegative women in order to determine if an intervention (educational intervention or vaccine) is effective. Efficacy would be measured by comparing the proportion of women who seroconvert in comparison groups (that is the proportion of women who become seropositive during the study). It is not possible to determine acquisition of infection by a different strain (re-infection) of CMV or reactivation of CMV in seropositive women using currently available techniques. Such intervention studies will need to enrol thousands of women and will be therefore require large amounts of resourcing, so being able to accurately power these studies is essential.

There is limited data on the seroprevalence of CMV amongst women of childbearing age in the UK.

Investigators will test stored antenatal serum from pregnant women from six sites across England. Investigators will test these samples at the point at which they would otherwise be destroyed, these samples would therefore not be utilised as part of clinical care. Investigators will not seek consent for testing of these samples from individuals and no results of blood tests will be provided to individuals. All pregnancies will be completed and therefore the result would have no impact on the antenatal care. There is no routine antenatal or postnatal screening done for CMV antibodies (to determine past of present infection) in the UK.

Samples will be fully anonymised within the University Hospital Southampton NHS Foundation Trust Specialist Virology Laboratory and tested in using routinely performed clinical procedures by NHS staff. No research staff will be involved in the transportation, receipt or testing of the samples. Results will be provided by NHS laboratory staff to researchers in fully anonymised form. Therefore at no time will researchers have access to patient identifiers on patient samples.

ELIGIBILITY:
Inclusion Criteria:

* Antenatal sera collected in the designated sites within the first 16 weeks of pregnancy and collected within a two-month period between 1st April 2019 and 1st October 2019 inclusive.

Exclusion Criteria:

* There are no exclusion criteria other than inability to fulfil the inclusion criteria above.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-05-03 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The seroprevalence of CMV in sera collected in the first trimester of pregnancy | 31/12/2021
  Proportion of samples that are CMV IgG+
The seroincidence of primary CMV infection in the first trimester of pregnancy | 31/12/2021
  Proportion of samples that are IgG+, IgM+ with low IgG avidity

IPD SHARING:
Plan to Share IPD: No
The study results will be published and IPD will be made available to researchers on reasonable request to the CI